CLINICAL TRIAL: NCT06591832
Title: Effect of Virtual Reality-Based Relaxation Exercise on Postoperative Pain and Kinesiophobia After Total Knee Replacement: Randomized Controlled Study
Brief Title: Effect of Virtual Reality-Based Relaxation Exercise on Postoperative Pain and Kinesiophobia After Total Knee Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aksaray University (Other)
Responsible Party: Principal Investigator, Zeynep Kocak, Principal Investigator, Aksaray University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/23-30
Record Dates: First submitted 2024-01-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-01

CONDITIONS: Randomized Controlled Trial
Keywords: Pain; kinesiophobia; virtual reality glasses
MeSH Terms: conditions — Pain; Kinesiophobia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Gorup (Experimental): Routine nursing practice will be performed and Virtual reality based progressive relaxation exercise will be applied
  Interventions: Other: Exercise
- Control Group (No Intervention): Routine nursing practice will be performed

INTERVENTIONS:
Other: Exercise — Virtual reality based progressive relaxation exercise
  Arms: Experimental Gorup

SUMMARY:
The aim of this study is to evaluate the effect of virtual reality-based relaxation exercise on pain and kinesiophobia in patients after total knee arthroplasty.

DETAILED DESCRIPTION:
Virtual reality application, which is a non-pharmacological application; It is a three-dimensional simulation model that gives individuals the feeling of reality and allows mutual communication with a dynamic environment created by computers, and studies determining the effects of the application are increasing day by day. Virtual reality-based rehabilitation is a promising approach to achieve recovery in many cases, optimize functional outcomes, and increase the clinical and social benefits of surgery . As a result, pain and fear of movement may negatively affect early functional results in patients undergoing total knee arthroplasty. Explaining how to change patients' fears, encouraging them to adopt positive attitudes and increasing their physical strength has an important place in determining the effectiveness of virtual reality application.

ELIGIBILITY:
Inclusion Criteria:

* The research included people between the ages of 40-75,
* Volunteering to participate in the research,
* Being able to understand and speak Turkish,
* Being able to understand the verbal, written and video explanations given,
* Having no problems communicating cognitively, affectively and verbally,
* Not having any obstacle to using virtual reality glasses,
* Patients who underwent unilateral TKA surgery,
* Using the SPH device at the same degree for three postoperative days after the FFP operation.
* Having the surgeon's permission

Exclusion Criteria:

* Patients who will undergo revision TDP surgery,
* Those who have a neurological disease that causes functional disability,
* Those with a diagnosed psychiatric disorder,
* Refusing to take the SPH device after the operation or taking it to a different degree,
* Those who have a condition that prevents them from wearing virtual glasses for any reason,
* These are patients after the FFP operation and outside the third postoperative day.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Min 0 Max 10 (As the score increases, the pain increases.)
  Visual Analog Scale
Tampa kinesiophobia scale | min 17 max 68 (As the score increases, the fear of movement increases.)
  assesses fear of movement

SECONDARY OUTCOMES:
After application Visual Analog Scale | Min 0 Max 10 (As the score increases, the pain increases.)
  Visual Analog Scale
After application Tampa kinesiophobia scale | min 17 max 68 (As the score increases, the fear of movement increases.)
  assesses fear of movement

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Koçak, Principal Investigator — Aksaray University; Funda Çetinkaya, Principal Investigator — Aksaray University
Locations (2):
- Turkey (Türkiye) (2):
  - Aksaray University, Aksaray
  - Aksaray Universitesi, Aksaray

IPD SHARING:
Plan to Share IPD: No